CLINICAL TRIAL: NCT04669223
Title: Clinical Efficacy and Complications of Small-bore Versus Ultra-small Bore Chest Drain in Malignant Pleural Effusion: a Randomized Clinical Trial
Brief Title: Comparing Different Sizes of Small-bore Chest Drains in Malignant Pleural Effusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult recruitment encountered during pandemic
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lui Mei Sze, Associate Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-582
Record Dates: First submitted 2020-12-01; First posted 2020-12-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2023-11

CONDITIONS: Pleural Effusion, Malignant; Lung Cancer Stage IV; Chest Tubes
MeSH Terms: conditions — Pleural Effusion, Malignant; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Seldinger chest drain 14F (Other): Patients with seldinger chest drain 14F inserted
  Interventions: Device: Seldinger chest drain insertion
- Seldinger chest drain 8F (Active Comparator): Patients with seldinger chest drain 8F inserted
  Interventions: Device: Seldinger chest drain insertion

INTERVENTIONS:
Device: Seldinger chest drain insertion — Different sizes of chest drain will be inserted with seldinger technique

SUMMARY:
Malignant pleural effusion (MPE) is a very common medical condition, especially among patients with disseminated cancers. Chest drain insertion aims to drain the pleural fluid collection and relieve dyspnea. Small bore chest tubes are recommended as the first line therapy for draining pleural effusions. However, there is no clinical data available to inform on the size of drains for better drainage. This is a randomized study comparing the two common bores of small bore chest drains in Hong Kong, and assess for its clinical efficacy and complication risks.

DETAILED DESCRIPTION:
Introduction: Malignant pleural effusion (MPE) is the commonest complication of lung cancer, and its associated symptoms are frequent causes of hospitalizations and morbidities in patients with disseminated cancers. Chest tube drainage is often performed for symptomatic relief. Recent clinical trials had shown that large-bore chest drains (>14 French) caused significantly more pain than smaller drain during the insertion procedure and when the drain was in situ, which prompts the shift of preference towards smaller chest drains in guideline and clinical practice. Chest drains as small-bore as 7-8 French have been used in many local centers for drainage of MPE, though little attention has been made to the possible higher occurrence of drain blockage, kinking or dislodgement before optimal effusion drainage is achieved, which may lead to a second procedure for drain replacement. Currently, there is no data informing the efficacy and complications of ultra-small chest drains in clinical use. Therefore, it is imperative to call for further research on the optimal size of the chest drain which can achieve satisfactory drainage and at the same time, of minimal complications.

Study design: Single-center, parallel group, single blinded, randomized controlled study Study site: Department of Medicine, Queen Mary Hospital Target study participants: Subjects with symptomatic MPE requiring chest drainage

Method and analysis: This randomized controlled study to compare the efficacy of ultra-small bore chest drains (8 Fr) with standard small bore chest drain (14 French) as the reference. Primary outcome is drain success defined by nearly complete drainage of MPE on chest radiograph on day 5 of the drain. Other secondary outcomes include pain according to the visual analogue scale, dyspnea relief and complications during the procedure and post - chest drain insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have cytologically/histologically proven pleural malignancy, or who have pleural effusion in the context of malignancy elsewhere
* The pleural effusion is at least moderate to massive and causes symptoms
* Ability to give informed written consent to the study

Exclusion Criteria:

* Age <18 years old
* Bleeding tendency not readily correctable (platelet < 100 x 10^9, INR ≥1.5 after transfusion)
* Hydropneumothorax before drain insertion
* Moderate-heavy septations in the pleural effusion (defined as a collection with more than 4 septations visible at the maximally septated area)
* Clinical emergency that an urgent chest drain is required
* Allergy to local anesthesia agents
* Blindness
* History of pleurodesis on the same side of malignant pleural effusion requiring drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with drainage success by day 5 of chest drain | Day 5 of chest drain insertion
  Drain success is defined by achieving nearly complete drainage through chest-x ray or ultrasound

SECONDARY OUTCOMES:
Pain assessed by visual analogue scale ( score from 1 to 10 )when drain is in-situ | Day 5 of chest drain insertion
  To record pain through visual analogue scale, which in higher score signifies worse pain
Change in dyspnea assessed by visual analogue scale for dyspnea ( score from 1 to 10 ) | Day 5 of chest drain insertion
  To record change in dyspnea through the dyspnea visual analogue scale, which a higher score signifies worse dyspnea
Rate of complications during and after insertion | Day 5 of chest drain insertion
  To record and analyse complications during and after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Mei Sze Macy Lui, MD, Principal Investigator — Associate Consultant
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Havelock T, Teoh R, Laws D, Gleeson F; BTS Pleural Disease Guideline Group. Pleural procedures and thoracic ultrasound: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii61-76. doi: 10.1136/thx.2010.137026. No abstract available. PMID 20696688
- [Background] Rahman NM, Pepperell J, Rehal S, Saba T, Tang A, Ali N, West A, Hettiarachchi G, Mukherjee D, Samuel J, Bentley A, Dowson L, Miles J, Ryan CF, Yoneda KY, Chauhan A, Corcoran JP, Psallidas I, Wrightson JM, Hallifax R, Davies HE, Lee YC, Dobson M, Hedley EL, Seaton D, Russell N, Chapman M, McFadyen BM, Shaw RA, Davies RJ, Maskell NA, Nunn AJ, Miller RF. Effect of Opioids vs NSAIDs and Larger vs Smaller Chest Tube Size on Pain Control and Pleurodesis Efficacy Among Patients With Malignant Pleural Effusion: The TIME1 Randomized Clinical Trial. JAMA. 2015 Dec 22-29;314(24):2641-53. doi: 10.1001/jama.2015.16840. PMID 26720026
- [Background] Parulekar W, Di Primio G, Matzinger F, Dennie C, Bociek G. Use of small-bore vs large-bore chest tubes for treatment of malignant pleural effusions. Chest. 2001 Jul;120(1):19-25. doi: 10.1378/chest.120.1.19. PMID 11451810
- [Background] Hallifax RJ, Psallidas I, Rahman NM. Chest Drain Size: the Debate Continues. Curr Pulmonol Rep. 2017;6(1):26-29. doi: 10.1007/s13665-017-0162-3. Epub 2017 Jan 26. PMID 28344925
- [Background] Mishra EK, Corcoran JP, Hallifax RJ, Stradling J, Maskell NA, Rahman NM. Defining the minimal important difference for the visual analogue scale assessing dyspnea in patients with malignant pleural effusions. PLoS One. 2015 Apr 15;10(4):e0123798. doi: 10.1371/journal.pone.0123798. eCollection 2015. PMID 25874452